CLINICAL TRIAL: NCT04255563
Title: Drug-coating Balloon Treatment in Coronary Artery Disease: a Prospective, Multicenter, Registry Study (ULTIMATE-DCB)
Brief Title: Drug-coating Balloon Treatment in Coronary Artery Disease
Acronym: ULTIMATE-DCB
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Junjie Zhang, Vice chief of the department of cardiology, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20200110-03
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCB treatment: DCB (Sequent® Please) treatment will be performed for suitable patients with CAD.
  Interventions: Device: DCB treatment

INTERVENTIONS:
Device: DCB treatment — DCB (Sequent® Please) treatment for CAD patients will be enrolled. Intravascular ultrasound (Boston Scientific®) guidance is recommended.

SUMMARY:
Drug-coated balloon (DCB) is an alternative choice for patients with coronary artery disease (CAD). This study is to investigate the efficacy and safety of DCB treatment in patients with CAD.

DETAILED DESCRIPTION:
This is a prospective, multi-center, registry to enroll patients undergoing DCB treatment.

All subjects undergoing DCB treatment will be enrolled in this study without strict inclusion and exclusion criteria. Data and images will be collected during the index procedure, and at the clinical and angiographic follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for DCB treatment

Exclusion Criteria:

* Pregnancy
* Contraindications to contrast media, antiplatelet therapy, or paclitaxel
* Expected life less than 12 months
* Cardiac shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with coronary artery disease undergoing DCB treatment will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
target vessel failure (TVF) at 12 months | 12 months
  TVF is defined as the composite of cardiac death, target-vessel myocardial infarction and ischemia-driven target- vessel revascularization.

SECONDARY OUTCOMES:
Parameter by quantitative coronary angiography at 7 months | 7 months
  Late lumen loss
Bleeding at 12 months | 12 months
  bleeding
Bailout drug-eluting stents (DES) implantation rate | During procedure
  Bailout DES implantation rate during procedure by angiographic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No